CLINICAL TRIAL: NCT00900536
Title: TRANSORCE (A Sub-study of SORCE)
Brief Title: DNA Analysis of Blood and/or Tissue Samples From Patients With Primary Kidney Cancer Receiving Sorafenib on Clinical Trial MRC-RE05-SORCE
Status: Completed | Type: Observational
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: MRC-RE05-TRANSORCE; CDR0000601175 (Registry Identifier: PDQ (Physician Data Query)); EU-20867; EUDRACT-2006-006079-19; ISRCTN38934710
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2008-11

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer; papillary renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Amplified Fragment Length Polymorphism Analysis; Immunohistochemistry

INTERVENTIONS:
Genetic: mutation analysis
Genetic: polymorphism analysis
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and/or tissue in the laboratory from patients with kidney cancer receiving sorafenib may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how well patients will respond to sorafenib.

PURPOSE: This research study is looking at the DNA in blood and/or tissue samples from patients with primary kidney cancer receiving sorafenib on clinical trial MRC-RE05-SORCE.

DETAILED DESCRIPTION:
OBJECTIVES:

* Examine the relationship between tumor genotype, expression, and patient outcome.
* Examine the relationship between constitutional genotype and patient outcome.

OUTLINE: This is a multicenter study.

Patients undergo blood and/or tissue sample collection for laboratory studies. Laboratory studies include generation of tissue microarrays; analysis of protein expression by immunohistochemistry; tumor DNA extraction and whole genome amplification; detection of VHL or other relevant gene mutations by direct sequencing; and constitutional (lymphocyte DNA) genotyping by single nucleotide polymorphism analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed resected renal cell carcinoma

  * Clear cell or non-clear cell tumor
* Receiving sorafenib tosylate on clinical trial MRC-RE05-SORCE

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-07; Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Relationship between tumor genotype, expression, and patient outcome
Relationship between constitutional genotype and patient outcome

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Eisen, Study Chair — Cancer Research UK
Locations (1):
- Addenbrooke's Hospital, Cambridge, England, United Kingdom